CLINICAL TRIAL: NCT00819273
Title: Investigation Into the CorrelAtion of pLasma Hs-CRP Concentrations and cardiovascuLar rISk in Korean populaTiOn
Acronym: CALLISTO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Hyunah Caroline, Choi / CV TA Physician, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CKR-DUM-2008/5
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: hsCRP
Keywords: hsCRP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients who have records of clinic visit with circulatory and endocrine internal medicines of nationwide tertiary hospitals within the last one year.

SUMMARY:
An observational, non-interventional, multi-centre study to provide further information on the utility of test for a predictive marker by investigating the current prevalence of high sensitivity CRP (hs-CRP) testing and characteristics of each CVD risk group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least one clinic visit record within the last 12 months from the date of data entry.
* Subjects with at least one hs-CRP level measured within the last 12 months from the date of data entry.

Exclusion Criteria:

* Use of statins or other lipid-lowering therapies including fibrates, niacin, and bile acid sequestrants in the past 3 months prior to hsCRP measurement
* Active inflammatory diseases documented during the period of CRP measurement
* Subjects taking immunosuppressants
* Findings of chronic inflammation: arthritis, lupus, or inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have records of clinic visit with circulatory and endocrine internal medicines of nationwide tertiary hospitals within the last one year.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Evaluate hs-CRP levels according to risk categories by the NCEP ATP III. | Within the last 12 months from the date of data entry.

SECONDARY OUTCOMES:
Evaluate a relationship between hs-CRP and each CHD CVD risk factor including LDL-C. | Within the last 12 months from the date of data entry.

CONTACTS AND LOCATIONS:
Overall Officials: Baek Sanghong, Ph.D., Principal Investigator — The Catholic University
Locations (10):
- South Korea (10):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Anyang-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Uijeongbu-si, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Jeonju
  - Research Site, Kwangju-si
  - Research Site, Seoul